CLINICAL TRIAL: NCT01807455
Title: An Open, Non-comparative Study of the Efficacy and Safety of Treatment of Acne Scars With Restylane Vital Lidocaine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05DF1206
Record Dates: First submitted 2013-03-06; First posted 2013-03-08 (Estimated); Results first posted 2016-01-25 (Estimated); Last update posted 2022-08-26 (Actual); Status verified 2015-12

CONDITIONS: Acne Scars

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Restylane Vital Lidocaine (Experimental)
  Interventions: Device: Restylane Vital Lidocaine

INTERVENTIONS:
Device: Restylane Vital Lidocaine

SUMMARY:
The purpose of this study is to demonstrate the efficacy and safety of Restylane Vital Lidocaine when acne scars are treated

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 25 to 45 years.
* Caucasian with Fitzpatrick skin type I-III.
* Must be cooperative and willing to comply with the instructions and procedures.
* Provision of signed and dated informed consent to participate in the study.
* Presence of depressed facial atrophic acne scars with a diameter of <4 mm according to at least SCAR-S score 3 category moderate (i.e. more than half of the face involved).

Exclusion Criteria:

* Icepick scarring or atrophic scars with a diameter of ≥4 mm covering more than 25% of the face.
* Active acne with inflammatory component.
* Post-surgical scars in the face.
* History of keloid formation or hypertrophic scars.
* Use of isotretinoin within 12 months of the baseline visit.
* Use of per oral or topical (facial) substances containing retinoids, bensoyl peroxide, alpha-hydroxy acid at a concentration above 10% or beta-hydroxy acid at a concentration above 2% or antibiotics within four months of the baseline visit.
* Concomitant anticoagulant therapy and therapy with inhibitors of platelet aggregation (e.g. aspirin or other nonsteroidal anti-inflammatory drugs [NSAIDs]), Omega-3 or vitamin E seven days before the injection, or a history of bleeding disorders.
* Use of anti-inflammatory agents seven days before the injection.
* History of radiation or skin tumours including actinic keratosis in the face.
* Active skin disease, inflammation or related conditions, such as infection, perioral dermatitis, seborrheic eczema and rosacea in the face.
* History of or active collagen diseases or autoimmune diseases such as systemic lupus erythematous, rheumatic arthritis, skin or systemic sclerosis.
* Previous hypersensitivity to HA.
* Previous hypersensitivity to lidocaine or other amide-type anaesthetics.
* Concomitant treatment with chemotherapy, immunosuppressive agents, immunomodulatory therapy (e.g. monoclonal antibodies), systemic or topical (facial) corticosteroids within 3 months of the baseline visit. (Inhaled corticoids are not an exclusion criterion).
* Presence of facial hair that may interfere with efficacy evaluations.
* Previous tissue augmenting therapy or revitalization treatment in the treatment area with HA or collagen, within 12 months of the baseline visit.
* Permanent implant or treatment with fillers based on other material than HA or collagen in the treatment area.
* Laser, e.g. carbon dioxide and Fraxel, dermabrasion or facial light therapy, e.g. IPL, in the treatment area within 12 months of the baseline visit.
* Chemical peeling in the treatment area within 6 months of the baseline visit.
* Previous surgery in the treatment area.
* Nicotine use within 6 months before the baseline visit.
* Pregnancy or breast feeding.
* Participation in any other clinical study within 30 days before inclusion.
* Any medical condition that in the opinion of the investigator makes the subject unsuitable for inclusion (e.g. severe chronic disease, epilepsy, impaired cardiac conduction, severely impaired hepatic function or severe renal dysfunction).
* Other condition preventing the subject from entering the study in the investigator's opinion, e.g. subjects not likely to avoid other facial cosmetic treatments, subjects anticipated to be unreliable or incapable of understanding the study assessment or unrealistic expectations of treatment result.
* Study staff or close relative of study staff (e.g. parents, children, siblings and spouse).

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2013-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Dierickx, MD, Principal Investigator
Locations (1):
- Skin and Laser Center, Boom, Belgium

RESULTS

PARTICIPANT FLOW:
Groups:
- Restylane Vital Lidocaine: Restylane Vital Lidocaine
Period: Overall Study
Arm/Group | Restylane Vital Lidocaine
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Restylane Vital Lidocaine
Number analyzed (Participants) | 12
Age, Continuous [Mean (Full Range); unit: years] | 33 [27 to 43]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of Acne Scarring and the Surrounding Skin Using the Global Aesthetic Improvement Scale
Description: Percentage of improved subjects at 36 weeks after first treatment session assessed using Subject GAIS. Scale range is Worse, No Change, Somewhat Improved, Much Improved and Very Much Improved. Alternatives Somewhat Improved to Very Much Improved are considered an improvement, i.e. a better outcome.
Time Frame: 36 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Restylane Vital Lidocaine
Number analyzed (Participants) | 12
percentage of participants | 100

2. Secondary Outcome: Evaluation of Skin Quality and Overall Satisfaction Using a Subject Satisfaction Questionnaire
Description: Percentage of subjects satisfied with the overall appearance of the face at 36 weeks after first treatment session. Scale range is Very dissatisfied, Somewhat dissatisfied, Neither satisfied nor dissatisfied, Somewhat satisfied and Very satisfied. Alternatives Somewhat satisfied to Very satified are considered a better outcome.
Time Frame: 36 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Restylane Vital Lidocaine
Number analyzed (Participants) | 12
percentage of participants | 83.3

3. Secondary Outcome: Evaluation of Acne Scarring Using the Scale for Acne Scar Severity (SCAR-S)
Description: Percentage of subjects improved at 36 weeks after first treatment session assessed using SCAR-S. Scale range is Very severe, Severe, Moderate, Mild, Almost clear and Clear. The alternative Clear is considered the best outcome. Improvement is considered to be at least one step improvement on the scale toward the alternative Clear.
Time Frame: 36 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Restylane Vital Lidocaine
Number analyzed (Participants) | 12
percentage of participants | 66.7

4. Secondary Outcome: Assessment of Local Tolerability After Treatment
Description: Number of subjects reporting anticipated injection-related reactions after treatment
Time Frame: 14 days
Measure: Number; unit: participants
Arm/Group | Restylane Vital Lidocaine
Number analyzed (Participants) | 12
participants | 12

5. Secondary Outcome: Adverse Event Reporting During the Study
Description: Number of subjects reporting at least one adverse event (assessed as unrelated or related to treatment)
Time Frame: 36 weeks
Measure: Number; unit: participants
Arm/Group | Restylane Vital Lidocaine
Number analyzed (Participants) | 12
participants | 8

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected by open questioning, information obtained from signs and symptoms detected during examination, observed by study personnel or spontaneous reports from the subjects.
Arm/Group | Restylane Vital Lidocaine
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 8/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Restylane Vital Lidocaine (N=12)
Implant site bruising (General disorders) | 2 (2)
Implant site erythema (General disorders) | 5 (8)
Implant site inflammation (General disorders) | 1 (1)
Implant site mass (General disorders) | 1 (1)
Implant site nodule (General disorders) | 5 (9)
Implant site pain (General disorders) | 2 (2)
Implant site swelling (General disorders) | 3 (3)
Injection site inflammation (General disorders) | 1 (1)
Injection site warmth (General disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other